CLINICAL TRIAL: NCT00578643
Title: HLA Matched Unrelated or Non-Genotype Identical Related Donor Transplantation For Chronic Granulomatous Disease
Brief Title: Matched Unrelated or Non-Genotype Identical Related Donor Transplantation For Chronic Granulomatous Disease
Acronym: MUNCHR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor, Hematology Oncology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14771-MUNCHR
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Chronic Granulomatous Disease
Keywords: Stem Cell Transplant; Chronic Granulomatous Disease; Fludarabine; Busulfan; Cyclophosphamide
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — Busulfan; Alemtuzumab; Cyclophosphamide; fludarabine; fludarabine phosphate; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic unrelated transplant (Experimental): Conditioning from Day -9 to Day -1. Stem cells given on Day 0. Busulfan, alemtuzumab, cyclophosphamide, fludarabine, cyclosporine, stem cell infusion.
  Interventions: Drug: Busulfan; Biological: Alemtuzumab; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Cyclosporine; Procedure: Stem Cell Infusion

INTERVENTIONS:
Drug: Busulfan — Days -9 through -6
  1 mg/kg initially (based on weight)
  Other Names: Busulfex
Biological: Alemtuzumab — Day -5 through Day -2
  Dose is based on weight:
  Less than 15 kg: 3 mg
  More than 15 kg to 30 kg: 5 mg
  More than 30 kg: 15 mg
  Other Names: Campath
Drug: Cyclophosphamide — Days -5 through -2
  50 mg/kg
  Other Names: Cytoxan
Drug: Fludarabine — Day -5 through Day -2
  30 mg/m^2
  Other Names: Fludara
Drug: Cyclosporine — Cyclosporine will be administered beginning Day -2. Initial dose will 5 mg/kg infused over 24 hours.
  Other Names: Sandimmune
Procedure: Stem Cell Infusion — Stem Cell: Either bone marrow, cord blood, or peripheral blood stem cells may be used for stem cell transplantation. It is desired to infuse: for bone marrow, nucleated cells ≥ 4 X 10^8/kg recipient weight; for cord blood ≥ 3 X 10^7/kg nucleated cells; for peripheral blood stem cells ≥ 1 X 10^/kg CD34+ cells.

SUMMARY:
This study is for patients with chronic granulomatous disease (CGD), which is a disorder of the immune system that puts them at risk for severe infections. CGD is caused by a genetic defect that stops or prevents the white blood cells from killing certain bacteria and fungi. This condition cannot presently be cured by standard treatment with drugs or surgery. Medicine including antibiotics, antifungals, and interferon gamma, may help some patients with CGD; however even with continuous treatment, most patients with CGD will have chronic and recurrent infections. Transfusion of white blood cells may help overcome infection, but white cell transfusions lead to allergic reactions and fever and the benefit of transfusion lasts only a matter of hours. Ultimately, chronic infections can damage or injure the body organs. Injury to the lung or liver can lead to lung or liver failure and death. Medicines used to treat infection can damage body organs too. Infections may become resistant to antibiotic or antifungal treatment, and infections not responding to treatment can be deadly.

It is now known that under specific conditions and with special treatment, blood stem cells (the cells that make blood) can be transplanted from one person to another. Stem cell transplantation has been done for patients with CGD who have a healthy sibling and who share the same immune type (HLA type) as the patient. Stem cell transplantation allows healthy or normal white cells from the stem cell donor to grow or develop in the patient's bone marrow. These healthy white cells can fight infection and prevent future infections for a patient with CGD.

Patients on this study will receive stem cells from a related or unrelated donor. The donor will be closely matched to the patient's immune type but the donor is not a sibling. The reason this treatment is investigational is that we do not know the likelihood of benefit that the patient will receive. It is possible that they will have great benefit, like some of the patients who have been transplanted from a brother or sister. It is possible that the side-effects of treatment may be too severe so that the transplant won't work.

The purpose of this research study is to evaluate whether or not patients with CGD treated with a stem cell transplant from a non-matched and/or non-related donor can have a good outcome from the procedure with an acceptable number of side-effects.

DETAILED DESCRIPTION:
In order to transplant stem cells we will need to give the patient drugs or high-dose chemotherapy to kill or destroy most of the blood forming and immune cells in the bone marrow. This is necessary to allow the donor stem cells to live and grow (engraft) in the bone marrow space. After the drug treatment is completed, the patient will be given the stem cells from the donor. The drug treatment is as follows:

Day -9 Busulfan

Day -8 Busulfan

Day -7 Busulfan

Day -6 Busulfan

Day -5 Alemtuzumab, Fludarabine, Cyclophosphamide

Day -4 Alemtuzumab, Fludarabine, Cyclophosphamide

Day -3 Alemtuzumab, Fludarabine, Cyclophosphamide

Day -2 Alemtuzumab, Fludarabine, Cyclosporine, Cyclophosphamide

Day -1 REST

Day 0 Stem cell infusion

The day after the chemotherapy treatment is completed, the patient will receive the healthy stem cells by vein, like a blood transfusion. Once in the bloodstream, the marrow cells will go to the bone marrow and grow.

It is also possible that if the marrow takes, it will cause a disease known as graft-versus-host disease (GVHD). To prevent GVHD, we will give the patient cyclosporine and Methotrexate. Methotrexate will be administered on Days 1, 3, 6 and 11 after the transplant. The cyclosporine therapy will continue for a longer period of time, however if the patient does not develop GVHD, it will be discontinued by 6 months after the stem cell transplant.

ELIGIBILITY:
INCLUSION CRITERIA:

CGD patients as documented by an abnormal NBT assay in a male patient and/or abnormal NADPH enzyme mutation confirmed by genetic analysis with abnormal NBT.

Patients must not have an HLA genotype identical donor.

Patients must have a 5/6 or 6/6 HLA-matched unrelated donor or a 5/6 or 6/6 HLA phenotype-matched related donor.

Patients must have had at least one serious infection characteristic of those manifested in patients with CGD.

Patients must not have active infection. An active infection may include the following: 1) clinical findings consistent with an infection such as fever, cavitary organ lesions, osteomyelitis; 2) progression of presumed infection based upon findings of diagnostic imaging (two or more studies at least 1 month a part).

No cumulative organ dysfunction that, in the estimation of the treating physicians, will diminish the patient's likelihood to survive this procedure.

Negative pregnancy test for post-pubertal female patients.

Echocardiogram shortening fraction >/= 28%.

DLCO 50% or greater predicted or FEV1 >/= 50% predicted.

EXCLUSION CRITERIA:

Active or uncontrolled infection (e.g. lung infection, cavitary organ lesions, osteomyelitis).

Markedly elevated C reactive protein or sedimentation rate relative to patient's baseline.

Invasive bone or bone marrow disease.

Lack of potential hematologic blood product donors in the past (related to McLeod phenotype).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-03; Primary Completion 2017-07-31 (Actual); Study Completion 2017-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krance, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Allogeneic Unrelated Transplant: Conditioning from Day -9 to Day -1. Stem cells given on Day 0. Busulfan, alemtuzumab, cyclophosphamide, fludarabine, cyclosporine, stem cell infusion.
  Busulfan: Days -9 through -6
  1 mg/kg initially (based on weight)
  Alemtuzumab: Day -5 through Day -2
  Dose is based on weight:
  Less than 15 kg: 3 mg
  More than 15 kg to 30 kg: 5 mg
  More than 30 kg: 15 mg
  Cyclophosphamide: Days -5 through -2
  50 mg/kg
  Fludarabine: Day -5 through Day -2
  30 mg/m^2
  Cyclosporine: Cyclosporine will be administered beginning Day -2. Initial dose will 5 mg/kg infused over 24 hours.
  Stem Cell Infusion: Stem Cell: Either bone marrow, cord blood, or peripheral blood stem cells may be used for stem cell transplantation. It is desired to infuse: for bone marrow, nucleated cells ≥ 4 X 10^8/kg recipient weight; for cord blood ≥ 3 X 10^7/kg nucleated cells; for peripheral blood stem cells ≥ 1 X 10^/kg CD34+ cells.
Period: Overall Study
Arm/Group | Allogeneic Unrelated Transplant
Started | 15
Completed | 13
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Analysis included 15 patients who underwent HLA matched unrelated or non-genotype identical related donor transplantation for chronic granulomatous disease(CGD).
Arm/Group | Allogeneic Unrelated Transplant
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6 [2 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 7
  Race/Ethnicity: Black or African American | 1
  Race/Ethnicity: Asian | 1
  Race/Ethnicity: Hispanic or Latino | 5
  Race/Ethnicity: Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Engraftment
Description: To estimate the engraftment rate for patients with CGD using busulfan, cyclophosphamide, fludarabine and alemtuzumab (Campath 1H) as conditioning therapy for SCT from 5/6 or 6/6 HLA-matched unrelated or 5/6 or 6/6 HLA phenotype-matched related donors.
Time Frame: 28 days post transplant
Measure: Number; unit: percentage of participants
Arm/Group | Allogeneic Unrelated Transplant
Number analyzed (Participants) | 15
percentage of participants | 100

2. Secondary Outcome: Number of Patients That Have Complete Donor Chimerism After Transplant.
Description: To estimate the likelihood of complete donor chimerism for patients with CGD using busulfan, cyclophosphamide, fludarabine and alemtuzumab (Campath 1H) as conditioning therapy for SCT from 5/6 or 6/6 HLA-matched unrelated or 5/6 or 6/6 HLA phenotype-matched related donors.
Time Frame: 120 days post transplant
Population: One patient died on day 62 post transplant and was not included in the analysis.
Measure: Number; unit: participants
Arm/Group | Allogeneic Unrelated Transplant
Number analyzed (Participants) | 14
participants | 13

3. Secondary Outcome: Number of Patients That Have Acute GVHD and Regimen Related Morbidity/Mortality Post Transplant.
Description: To estimate the risk for acute GVHD and regimen related morbidity/mortality for patients with CGD following stem cell transplant from 5/6 or 6/6 HLA matched unrelated or 5/6 or 6/6 HLA phenotype matched related donors.
Time Frame: Assessed between day 0 and day 100 post transplant
Population: One patient who died on day 62 post transplant without developing acute GVHD was not assessed for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Unrelated Transplant
Number analyzed (Participants) | 14
Participants
  None | 8
  Grade I | 6
  Grade II | 0
  Grade III-IV | 0

4. Secondary Outcome: Number of Patients That Have Chronic GVHD and Regimen Related Morbidity/Mortality Post Transplant.
Description: To estimate the risk for chronic GVHD and regimen related morbidity/mortality for patients with CGD following stem cell transplant from 5/6 or 6/6 HLA matched unrelated or 5/6 or 6/6 HLA phenotype matched related donors.
Time Frame: Assessed between day 100 and day 365 post transplant
Population: One patient died on day 62 post transplant, and one patient was lost to F/U on day 163 post transplant. They were not assessed for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Unrelated Transplant
Number analyzed (Participants) | 13
Participants
  Yes | 0
  No | 13

ADVERSE EVENTS:
Time Frame: Adverse events excluding fevers and hematological toxicities were collected up to 30 days after transplant. SAEs excluding fevers and hematological toxicities were collected up to 100 days after transplant.
Description: An adverse event was defined as grade III or grade IV toxicity by the NCI Common Toxicity Criteria Version 3.0. A SAE is any adverse event that was fatal, life threatening , required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product(s) or considered a significant medical event by the investigator.
Arm/Group | Allogeneic Unrelated Transplant
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Unrelated Transplant (N=15)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Constitutional Symptoms - Other: Multiorgan failure (General disorders) | 1 (1)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1 (1)
Gastrointestinal-Other: Eosinofilic enteritis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Hematuria (in the absence of vaginal bleeding) (Infections and infestations) | 1 (1)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e (Infections and infestations) | 1 (2)
Infection without neutropenia (Infections and infestations) | 1 (1)
Infection - Other: Adenovirus viremia, BK viruria, CMV viremia (Infections and infestations) | 1 (1)
Infection - Other: Hemorrhagic cystitis with BK virus, adenovirus, and CMV (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 1 (1)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Pleural effusion (non-malignant) 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other: Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Unrelated Transplant (N=15)
Hypertension (Cardiac disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1 (3)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 1 (1)
Hematuria (in the absence of vaginal bleeding) (Infections and infestations) | 1 (1)
GGT (Gamma-Glutamyl transpeptidase) (Hepatobiliary disorders) | 2 (3)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 2 (2)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 1 (1)
Catheter-related infection (Infections and infestations) | 1 (1)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia(ANC<1.0x10e9/L) (Infections and infestations) | 3 (3)
Infection without neutropenia (Infections and infestations) | 2 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 5 (6)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (2)
Amylase (Metabolism and nutrition disorders) | 1 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Lipase (Metabolism and nutrition disorders) | 1 (1)
Seizure(s) (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT00578643/Prot_SAP_000.pdf